CLINICAL TRIAL: NCT00787306
Title: Multidisciplinary Cardiovascular Health And Risk Modification in Family Health Teams
Brief Title: Cardiovascular Health And Risk Modification in Family Health Teams
Acronym: Multi-CHARM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Warren McIsaac, Associate Professor, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MOH-1048
Record Dates: First submitted 2008-11-06; First posted 2008-11-07 (Estimated); Last update posted 2018-04-03 (Actual); Status verified 2018-03

CONDITIONS: Cardiovascular Risk Factors; Hypertension; Hyperlipidemia; Diabetes
Keywords: chronic disease management; decision aids; cardiovascular risk factors
MeSH Terms: conditions — Hypertension; Hyperlipidemias; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Multi-faceted Cardiovascular Decision Support (Experimental): Risk factor active surveillance, multi-disciplinary disease management and decision aid intervention
  Interventions: Behavioral: Active risk factor surveillance
- Control Usual Care (Other): Usual care in a wait-list control arm that receives the experimental intervention after 6 months.
  Interventions: Behavioral: Active risk factor surveillance

INTERVENTIONS:
Behavioral: Active risk factor surveillance — Cardiovascular risk status assessment followed by active surveillance and physician review where risk factor control is suboptimal

SUMMARY:
Cardiovascular diseases remain the main cause of mortality in Canada. While effective interventions are available for reducing the risk of cardiovascular disease,there continue to be gaps between the potential reduction in risk that could be achieved by effectively managing these risk factors and levels of risk factor control currently in clinical practice. This study will evaluate the ability of a different model of risk factor care using other health providers assisting family doctors, along with information aids for patients and health professionals,to achieve better levels of cardiovascular risk factor control in adults.

ELIGIBILITY:
Inclusion Criteria:

* adults 50 to 80 years of age
* having attending a family medicine clinic for more than one year

Exclusion Criteria:

* not able to participate for one year
* not able to read English
* requires house calls
* nursing home resident
* cognitive impairment
* current chest pain or symptoms of active coronary heart disease

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 229 (Actual)
Dates: Start 2008-10; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
mean systolic blood pressure | 6 months

SECONDARY OUTCOMES:
Proportion of adults with 3 cardiovascular risk factors under optimal control | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Warren J McIsaac, MD, Principal Investigator — Granovsky Gluskin Family Medicine Centre, Mount Sinai Hospital
Locations (1):
- Granovsky Gluskin Family Medicine Cwntre, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No